CLINICAL TRIAL: NCT05596942
Title: Evaluating the Efficacy of Channa Striata in Stabilizing eNOS in Patients With Septic: A Randomized Control Trial.
Brief Title: Evaluating the Efficacy of Channa Striata in Stabilizing eNOS in Patients With Septic.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Septian Adi Permana, Intensivist, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Septian Adi P
Record Dates: First submitted 2022-09-22; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Sepsis
Keywords: sepsis; eNOS; NLR; PLR; Channa striata; albumin; inflammation; anti-oxidant
MeSH Terms: conditions — Sepsis; Inflammation | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albumin Chana Striata Extract (Experimental)
  Interventions: Dietary Supplement: Albumin Channa Striata Extract
- Human Albumin (Active Comparator)
  Interventions: Dietary Supplement: Albumin Channa Striata Extract

INTERVENTIONS:
Dietary Supplement: Albumin Channa Striata Extract — This study is a randomized controlled trial of 42 patients at the ICU of Dr. Moewardi General Hospital. The control group received 20 grams of human albumin on the first day and the study group received 15 grams of Channa striata extract daily for two days. Subsequently, eNOS, NLR and PLR are measured before and three days after treatment, and the examiners compare the three markers statistically.
  Other Names: Human Albumin

SUMMARY:
Sepsis is an inflammation response produced by the host's immune system, which is agrravated by oxidative stress. One of the adjuvant therapy according to Surviving Sepsis Campaign Guideline is albumin, which has anti-inflammatory and anti-oxidant effects. However, human albumin is quite expensive, and other forms with similar potency and less costs are needed, one of which is Channa striata extract. Therefore, this study is conducted to compare albumin and human albumin, specifically their anti- inflammatory and anti-oxidant properties by assessing the eNOS marker, neutrophil/lymphocyte ratio (NLR) and platelet/lymphocyte ratio (PLR) in patient with sepsis.

DETAILED DESCRIPTION:
In summary, this study showed that Channa striata extract has a better outcome in stabilizing eNOS level in patient with sepsis than human albumin 20%, and it has a potential benefit in stabilizing NLR values. However, further studies with a larger sample and a more advanced phase of sepsis are needed.

ELIGIBILITY:
Inclusion Criteria:

* patients sepsis who met the qSOFA criteria ≧ 2 [two of which: unconsciousness (Glasgow Coma Scale ≤14)
* respiratory rate > 22 and systolic blood pressure ≤ 100 mmHg],
* aged ≧ 18 years
* admitted to intensive care unit and high care unit at Dr. Moewardi General Hospital

Exclusion Criteria:

* patients with severe trauma
* blood loss in stage three or higher
* stress ulcers
* a history of nephrotic syndrome
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Endothelial Nitric Oxide Synthase | three days after treatment
  Measured before and three days after treatment, and the examiners compare the three markers statistically.

SECONDARY OUTCOMES:
Neutrophil-Lymphocyte Ratio | three days after treatment
  Measured before and three days after treatment, and the examiners compare the three markers statistically
Platelet-Lymphocyte Ratio | three days after treatment
  Measured before and three days after treatment, and the examiners compare the three markers statistically

CONTACTS AND LOCATIONS:
Locations (1):
- Moewardi General Hospital, Sukoharjo, Central Jave, Indonesia

IPD SHARING:
Plan to Share IPD: Yes